CLINICAL TRIAL: NCT02271724
Title: sCD163 & CD19 as Candidate Biomarkers in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) - A Study of sCD163 in the Cerebrospinal Fluid
Brief Title: sCD163 & CD19 as Candidate Biomarkers in CIDP and MMN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CIDP CD163; 1-10-72-300-14 (Other: The National Committee on Health Research Ethics (Denmark))
Record Dates: First submitted 2014-10-09; First posted 2014-10-22 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2015-09

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: CIDP; MMN; Spinal fluid; CD163; CD19
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Spinal fluid and blood sample for identification of different factors
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- CIDP/MMN newly diagnosed (drug naive): Patients, who are suspected to suffer from CIDP or MMN, will undergo a lumbar puncture as a part of the diagnostic procedure. We expect to include 5-10 patients.
  Lumbar puncture Blood sample
  Interventions: Procedure: Lumbar puncture; Procedure: Blood sample
- CIDP/MMN treated: All patients with established CIDP in maintenance treatment with SCIG or IVIG are recruited from local registries at the outpatient clinic at Department of Neurology, Aarhus University Hospital.
  We expect that 10-15 patients with CIDP and MMN treated with SCIG or IVIG eligible for inclusion. Furthermore, we expect to include 10 CIDP and MMN patients in maintenance therapy from the outpatient clinics at Department of Neurology, Odense University Hospital and Department of Neurology, Aalborg University Hospital.
  Interventions: Procedure: Lumbar puncture; Procedure: Blood sample
- Other peripheral neuropathies: Patients who are diagnosed with other causes of peripheral neuropathies than CIDP. We expect to include 20 patients
  Interventions: Procedure: Lumbar puncture; Procedure: Blood sample
- Syptomatic controls: Controls include patients with unspecified neurological symptoms or diseases who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work up irrespective of this study plus healthy controls. We expected to include 40-50 symptomatic controls
  Interventions: Procedure: Lumbar puncture; Procedure: Blood sample

INTERVENTIONS:
Procedure: Lumbar puncture — Lumbar puncture for spinal fluid
  Other Names: Spinal tap
Procedure: Blood sample — Blood sample

SUMMARY:
Chronic inflammatory demyelinating polyneuropathy (CIDP) and multifocal motor neuropathy (MMN) are characterized by progressive deterioration in muscle strength, loss of sensibility, diminished or absent reflexes and impaired fine motor control. Often it is caused by demyelination which is suitable for treatment but damage to the axons may also occur especially in case of insufficient treatment.

CIDP and MMN are immune mediated neuropathies in which first choice of treatment is intravenous immunoglobulin (IVIG), although the mechanisms underlying the effect of the IVIG is not yet clarified.

The patients are diagnosed by electrophysiological examination and elevated level of protein in the cerebrospinal fluid. The diagnosis may be difficult to make due to great clinical variation and insensitive examinations methods including lack of biomarkers.

The purpose of this study is to define if patients treated with SCIG and IVIG for CIDP and MMN have higher concentrations of sCD163 and CD19 in their cerebrospinal fluid and serum compared with symptomatic control subjects and is related to disease severity. Furthermore it is to define if patients newly diagnosed with CIDP or MMN have higher levels of sCD163 and CD19, than patients treated regularly with SCIG and IVIG.

DETAILED DESCRIPTION:
Chronic inflammatory peripheral neuropathies are characterized by progressive deterioration in muscle strength, loss of sensibility, diminished or absent reflexes and impaired fine motor control. Often it is caused by demyelination which is suitable for treatment but damage to the axons may also occur especially in case of insufficient treatment. Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) and multifocal motor neuropathy (MMN) are diagnosed by electrophysiological examination, which shows signs of demyelination and conduction blocks. Moreover, in CIDP an elevated level of protein in the cerebrospinal fluid and in MMN detection of anti-GM1 antibodies in the blood support the diagnosis.

The patients suffer from a disabling diffuse weakness of the muscles. The diagnosis primarily relies on the neurophysiological examination and, however, the diagnosis may be difficult to make due to great clinical variation and insensitive examinations methods including lack of biomarkers.

Treatment of CIDP and MMN CIDP and MMN are immune mediated neuropathies in which first choice of treatment is intravenous immunoglobulin (IVIG), although the mechanisms underlying the effect of the IVIG is not yet clarified.

Previous study implies that Fc receptors on natural killer cells is the target for IVIG, because the cytotoxic activity of NK cells was suppressed, partly caused by a dose-dependent decline in the number of circulating NK cells. Furthermore, a dose-dependent blockage of CD16 was present.

Subcutaneous administration of immunoglobulins (SCIG) has been studied as an alternative route to IVIG in CIDP and MMN. The conclusion was that SCIG is feasible, safe and effective. Thus SCIG improved muscle strength, walking performance and disability score compared to placebo and IVIG. SCIG has only local side effects compared to IVIG and furthermore the majority of patients preferred SCIG to IVIG, because of autonomy and maintenance of stable levels of muscle performance.

It is well known that around 30% of CIDP patients over year no longer need treatment to maintain muscle strength. Immunoglobulin treatment is costly and may, when administrated intravenously, induce severe side effects (e.g. thromboembolism, hemolytic anemia and exfoliative dermatitis). Therefore only patients that clearly respond should be treated. On the other hand, it is important to treat in time to reduce morbidity and disability.

Present examination methods Patients suspected for CIDP or MMN will be diagnosed based on the medical history, clinical examinations and neurophysiological findings. However, the diagnosis includes a plethora of criteria, which illustrates the difficulty of developing exact standards for CIDP and MMN that may have variable clinical presentations.

Furthermore, as described earlier electrophysiological examination is recommended for all patients suspected for CIDP or MMN. The electrophysiological criteria consist of partial conduction block, conduction velocity slowing, dispersion and distance dependent reduction of compound motor action potential amplitude. As for the medical history and clinical examinations, the electrophysiological examination is not always conclusive. The Koski criteria and the criteria from EFNS /PNS are two different sets of criteria, which are frequently used. Even so it is important to keep in mind that the Koski criteria have a sensitivity and specificity of 63 and 99 percent, whereas the EFNS had a sensitivity and specificity of 81 and 97 percent. In addition to this, early treatment for CIDP has made the progression more difficult to characterize as a temporal component has been changed.

It is still controversial whether CIDP and MMN are specific disease entities or rather syndromes. MMN is in many ways similar to CIDP but as opposed to CIDP MMN is characterized by no sensory disturbance, slower progression and with asymmetric presentation.

The specific causes of the diseases are still unknown but it is generally accepted that the pathologies of CIDP and MMN are immunologically based with multiple triggers. According to this theory both the cellular and the humoral part of the immune system is involved.

Several inflammatory biomarkers have been studied in relation to CIDP Including cytokines in CSF. The study measured Interleukin (IL)-12 and IL-15 (the major growth and differentiation factors for Th-1 cells) and IL-17 (a marker of Th-17 cell expansion and activation). Especially IL-12 was found to be involved as potential marker of immune activation in CIDP.

Nerve biopsy has also been used in search of in situ biomarkers. The conclusion was that even though the total numbers of inflammatory cells did not distinguish well between CIDP and non-inflammatory neuropathies, the pattern of macrophage clusters around endoneurial vessels could be a simple marker of inflammation with good sensitivity and specificity.

Furthermore, another study has found that CIDP is associated with a high level of haptoglobin in the CSF. The underlying mechanisms behind this has not yet been clarified. Nevertheless, this opens for haptoglobin as a possible useful biomarker.

Cluster of differentiation 19 (CD-19)- a promising B cell target! A study on spontaneous autoimmune polyneuropathy (SAP) in B7-2 knock- out non-obese diabetes mice, which is an animal model and mimics the chronic progressive form of human CIDP, has showed that treatment with anti-CD19 monoclonal antibody (mAb) results in depletion of B-cells and plasmablasts accompanied by decreased serum IgG and IgM levels and depletion of P0-specific plasmablasts and B-cells. CD-19 is a protein found on the surface of normal and neoplastic B-cells, from the early pre-B cell stage of development through to the early stages of plasma cell differentiation. The majority of B-cell lineage malignancies express CD19 at high levels. Therefore, CD19 is a broad marker of the B-cell lineage and represents a potentially important target for unconjugated mAb immunoteraphy. In another study by stimulating the CD19 B cell isolated from blood samples of CIDP patients, the B-cell immunoreactivity was enhanced but within 3 days of IVIG infusions, the B-cell level in CIDP was downregulated.

Cluster of differentiation 163 (CD-163) - a new way to measure CIDP and MMN? CD-163 is a scavenger receptor (recognizes and uptakes macromolecules) which marks the monocyte-macrophage activation. CD163 works for macrophages as a receptor for hemoglobin-haptoglobin complexes. The soluble form of the receptor is called sCD163 and is found in plasma, where it is found to be up regulated in a large range of inflammatory diseases.

Values which is Increased strongly (>20mg/l) is seen in diseases like macrophage activating syndrome, haemophagocytic syndrome and acute hepatic failure. Furthermore, the level of sCD163 reflects the activity of the disease. Patients with increasing and high values are found to have unfavorable prognosis. Increased values (5-20 mg/l) are seen in hepatic disease, sepsis and Gaucher's disease. Septic patients with values greater than 10 mg/l have a 10 times greater risk of fatal outcome. Values which is slightly increased (3-5 mg/l) is often seen in inflammatory of infectious conditions and in cancer.

Hypothesis Patients treated with SCIG for CIDP and MMN have higher concentrations of sCD163 and CD19 in their cerebrospinal fluid and serum compared with healthy control subjects and is related to disease severity.

Patients newly diagnosed with CIDP or MMN have higher levels of sCD163 and CD19, than patients treated regularly with SCIG.

Purpose To define the concentration of sCD163 and CD19 in the cerebrospinal fluid and serum in patients with CIDP or MMN compared with controls (patients with unspecified neurological symptoms or disease).

Method Data Sources Data used in this study will originate from several sources, such as the Danish Civil Registration Registry, the Danish National Patient Registry and the Danish national prescription registry.

Information from the medical record will be included and used in this project including past medical history, actual use of drugs, results of biochemical analyses and brain imaging, abnormalities at the clinical examinations and the conclusions from the doctors diagnostic workup.

Study population

The study population will consist of four subgroups:

Recruitment All participants will receive information about the project and will be asked to give their content to participation.

Participants will receive written and oral information about the study. The oral information will take place at Department of Neurology, Aarhus Universitetshospital. Moreover, the pamphlet " Før du deltager i et sundhedsvidenskabeligt forsøg"(about participating in a clinical trial) will be handed out.

The information will be given by consultant Henning Andersen, MD Lars Makrvardsen or stud. med Malalai Musleh . It is possible for the participants to bring a companion and they are offered one week to consider the participation.

Access to patient records will be requested, which will be provided in the written information material.

If new knowledge about disadvantages of participating in the study appears the participants will be informed immediately. Moreover, the participant will be informed if evaluations during the study bring knowledge about the general health status of the patient, unless this has been clearly rejected by the patient.

By the end of the study it is possible for participants to contact the study coordinator to get information about study results.

Participants will not receive any form of payment, but can receive compensation for transportation The participation implies extraction 3-5 ml of spinal fluid and a blood sample about 10 ml, which will be used for analysis of certain biomarkers, such as sCD163, CD19 and myelin proteins.

Other examination

Patients with CIDP and treatment with SCIG or IVIG plus drug-naïve CIDP patients will undergo a clinical examination with the following:

* Neuropathy Impairment Score (NIS)
* Overall Disability Sum Score (ODSS)
* Neuropathy Symptom Score (NSS) Disorders or treatments that contraindicate a lumbar puncture. In case an included patient turn out to meet the exclusion criteria after analyses of the spinal fluid, the patient will be replaced by a new patient.

At all times during the diagnostic work-up and consequently in the research project the investigators will do this with respect for the patients mental and physical condition. The research project will be carried out according to the Act on Processing of Personal Data and, furthermore, the project will be submitted to the common regional information system for Region Midtjylland.

Analyses The spinal fluid and the serum will be analysed at the Department of Clinical Medicine, Aarhus University Hospital. The spinal fluid and blood samples will be deposited in a research biobank at Aarhus University Hospital. The plan is to carry out all the biochemical analyses at the same time when all samples are collected. In the end of the project, the samples will be pseudo anonymised. Any excess biological material will be transferred to a biobank for future research.

The concentrations of sCD163 in spinal fluid and serum will be analyzed by already established techniques at the Department of Clinical Medicine, Aarhus University Hospital.

The concentrations of CD19 in spinal fluid and serum will be analyzed by established techniques at the Department of Immunology, Aarhus University Hospital.

Power and Statistical analyses Because of the rareness of both CIDP and MMN and the few number of patients it is not relevant to make Power calculations.

The program STATA will be used for statistical analyses. Parametric or non-parametric tests will be used depending of the normal distribution of data. In all statistical analysis a 5% level of significance will be used.

Perspectives Due to the many clinical variants of inflammatory polyneuropathies and due to the lack of biomarkers, it remains difficult to diagnose CIDP. It is very important to identify new methods for diagnosis and monitoring of patients with CIDP. This may also enable better prediction of the prognosis and the level of treatment needed.

The pathology of CIDP is still unknown but it is known to be immune mediated. In several studies sCD163 has been shown to up regulated in a larger range of inflammatory diseases suggesting sCD163 to be a relevant biomarker for CIDP.

It has also been proved that CD19 is a promising B-cell target for the development of disease-modifying agents in autoimmune neuropathies.

These findings can be used as diagnostic markers in patients with CIDP and MMN. Ethical considerations All the participants will be informed orally and in writing about the study and will receive consideration with a view to whether they want to participate. Signed consent will be given.

The tests performed on the patients involved in this research project are lumbar puncture, blood sampling and clinical examination.

A lumbar puncture is a procedure used to collect cerebral spinal fluid (CSF) for analysis. CSF is a promising source of biomarkers in CIDP since the proximal nerve roots, which are affected early in the disease, are in close anatomical contact with the CSF space. During the procedure a hollow needle is used to penetrate the spinal canal at the level of the third- to-fourth or fourth-to-fifth lumbar vertebra in the low back. CSF then drips out through the needle and is collected. It involves some risk to perform a lumbar puncture, which include post lumbar puncture headache with an incidence of 12%, most common in younger patients. Most frequently, the headache has a short duration and it may be cured with application of a blood -patch. Moreover, lumbar puncture can cause temporary lumbar pain and an accumulation of blood underneath the skin. There is a very low risk of bleeding in the epidural space with compression of spinal nerves and an even lower risk of infections (meningitis or meningoencephalitis).

However, it is important to highlight that lumbar puncture is part of routine diagnostic workout for neuropathy. However, CIDP patients treated with SCIG or IVIG will have a lumbar puncture for research purposes only. There are no further risks associated with collection of an extra sample of spinal fluid or blood. In consideration of the low risk involved in this project, the seriousness and costs of the disease and the potential to identify a relevant biomarker in CIDP, we consider this project to be ethically acceptable.

Publication Positive, negative as well as inconclusive results from this study will be published. The results will be written in an article for publication in an English written peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CIDP or MMN or patients suspected to have CIDP or MMN

Controls:

* Age >18 years

Exclusion Criteria:

* <18 years
* Acute infections including neuroinfection
* Diabetes
* Other disorders known to have elevated levels of sCD163 and CD19
* Disorders or treatments that contraindicate a lumbar puncture.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with CIDP and MMN in maintenance treatment with SCIG or IVIG
  * Patients with newly diagnosed CIDP and MMN (drug-naïve)
  * Patients with other causes of peripheral neuropathies
  * Symptomatic controls
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Concentrations of sCD-163 and CD19 in patients with CIDP and MMN. | Day 1

SECONDARY OUTCOMES:
Concentration of sCD163 and CD19 in newly diagnosed compared with established CIDP and MMN | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Principal Investigator — Department of Neurology, Aarhus University Hospital
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Background] Bohn AB, Nederby L, Harbo T, Skovbo A, Vorup-Jensen T, Krog J, Jakobsen J, Hokland ME. The effect of IgG levels on the number of natural killer cells and their Fc receptors in chronic inflammatory demyelinating polyradiculoneuropathy. Eur J Neurol. 2011 Jun;18(6):919-24. doi: 10.1111/j.1468-1331.2010.03333.x. Epub 2011 Jan 11. PMID 21219545
- [Background] Markvardsen LH, Debost JC, Harbo T, Sindrup SH, Andersen H, Christiansen I, Otto M, Olsen NK, Lassen LL, Jakobsen J; Danish CIDP and MMN Study Group. Subcutaneous immunoglobulin in responders to intravenous therapy with chronic inflammatory demyelinating polyradiculoneuropathy. Eur J Neurol. 2013 May;20(5):836-42. doi: 10.1111/ene.12080. Epub 2013 Jan 7. PMID 23294032
- [Background] Harbo T, Andersen H, Hess A, Hansen K, Sindrup SH, Jakobsen J. Subcutaneous versus intravenous immunoglobulin in multifocal motor neuropathy: a randomized, single-blinded cross-over trial. Eur J Neurol. 2009 May;16(5):631-8. doi: 10.1111/j.1468-1331.2009.02568.x. Epub 2009 Feb 19. PMID 19236457
- [Background] Van den Bergh PY, Pieret F. Electrodiagnostic criteria for acute and chronic inflammatory demyelinating polyradiculoneuropathy. Muscle Nerve. 2004 Apr;29(4):565-74. doi: 10.1002/mus.20022. PMID 15052622
- [Background] Harbo T, Andersen H, Jakobsen J. Acute motor response following a single IVIG treatment course in chronic inflammatory demyelinating polyneuropathy. Muscle Nerve. 2009 Apr;39(4):439-47. doi: 10.1002/mus.21305. PMID 19229876
- [Background] Markvardsen LH, Jakobsen J. [Exfoliative dermatitis as a side effect of intravenous immunoglobulin treatment]. Ugeskr Laeger. 2011 Oct 24;173(43):2725-6. Danish. PMID 22027232
- [Background] Markvardsen LH, Christiansen I, Harbo T, Jakobsen J. Hemolytic anemia following high dose intravenous immunoglobulin in patients with chronic neurological disorders. Eur J Neurol. 2014;21(1):147-52. doi: 10.1111/ene.12287. Epub 2013 Nov 4. PMID 24180709
- [Background] Fuglsang-Frederiksen A, Pugdahl K. Current status on electrodiagnostic standards and guidelines in neuromuscular disorders. Clin Neurophysiol. 2011 Mar;122(3):440-455. doi: 10.1016/j.clinph.2010.06.025. Epub 2010 Jul 31. PMID 20673740
- [Background] Rentzos M, Angeli AV, Rombos A, Kyrozis A, Nikolaou C, Zouvelou V, Dimitriou A, Zoga M, Evangelopoulos ME, Tsatsi A, Tsoutsou A, Evdokimidis I. Proinflammatory cytokines in serum and cerebrospinal fluid of CIDP patients. Neurol Res. 2012 Nov;34(9):842-6. doi: 10.1179/1743132812Y.0000000074. Epub 2012 Sep 4. PMID 22947427
- [Background] Stubgen JP. A review of the use of biological agents for chronic inflammatory demyelinating polyradiculoneuropathy. J Neurol Sci. 2013 Mar 15;326(1-2):1-9. doi: 10.1016/j.jns.2013.01.003. Epub 2013 Jan 19. PMID 23337197
- [Background] Sommer C, Toyka K. Nerve biopsy in chronic inflammatory neuropathies: in situ biomarkers. J Peripher Nerv Syst. 2011 Jun;16 Suppl 1:24-9. doi: 10.1111/j.1529-8027.2011.00301.x. PMID 21696493
- [Background] Zhang HL, Zhang XM, Mao XJ, Deng H, Li HF, Press R, Fredrikson S, Zhu J. Altered cerebrospinal fluid index of prealbumin, fibrinogen, and haptoglobin in patients with Guillain-Barre syndrome and chronic inflammatory demyelinating polyneuropathy. Acta Neurol Scand. 2012 Feb;125(2):129-35. doi: 10.1111/j.1600-0404.2011.01511.x. Epub 2011 Mar 24. PMID 21434877
- [Background] Kjaergaard AG, Rodgaard-Hansen S, Dige A, Krog J, Moller HJ, Tonnesen E. Monocyte expression and soluble levels of the haemoglobin receptor (CD163/sCD163) and the mannose receptor (MR/sMR) in septic and critically ill non-septic ICU patients. PLoS One. 2014 Mar 17;9(3):e92331. doi: 10.1371/journal.pone.0092331. eCollection 2014. PMID 24637679
- [Background] Etzerodt A, Moestrup SK. CD163 and inflammation: biological, diagnostic, and therapeutic aspects. Antioxid Redox Signal. 2013 Jun 10;18(17):2352-63. doi: 10.1089/ars.2012.4834. Epub 2012 Oct 19. PMID 22900885
- [Background] Moller HJ. Soluble CD163. Scand J Clin Lab Invest. 2012 Feb;72(1):1-13. doi: 10.3109/00365513.2011.626868. Epub 2011 Nov 7. PMID 22060747
- [Background] Abraham PM, Quan SH, Dukala D, Soliven B. CD19 as a therapeutic target in a spontaneous autoimmune polyneuropathy. Clin Exp Immunol. 2014 Feb;175(2):181-91. doi: 10.1111/cei.12215. PMID 24116957
- [Background] Korporal-Kuhnke M, Haas J, Schwarz A, Jarius S, Wildemann B. Plasmacytosis is a common immune signature in patients with MMN and CIDP and responds to treatment with IVIg. J Neuroimmunol. 2015 Jan 15;278:60-8. doi: 10.1016/j.jneuroim.2014.11.012. Epub 2014 Nov 22. PMID 25595253
- See also: Chronic inflammatory demyelinating polyneuropathy: Etiology, clinical features, and diagnosis — http://uptodate.com/contents/chronic-inflammatory-demyelinating-polyneuropathy-etiology-clinical-features-and-diagnosis